CLINICAL TRIAL: NCT06844019
Title: Birth & Breastfeeding Support Study
Acronym: BABSS
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Hanna Jangö, Associate Professor, Consultant Obstetrician, PhD, University of Copenhagen
Other Study IDs: F-24074649
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Breastfeeding; Breastfeeding Initiation; Breastfeeding Duration; Birth; Birth Practices; Gestational Diabetes Mellitus (GDM); Preeclampsia
Keywords: Birth, birth practices, gestational diabetes, preeclampsia; breastfeeding
MeSH Terms: conditions — Breast Feeding; Diabetes, Gestational; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cesarean Section: Birth by cesarean section and exclusive breastfeeding at 3 months of age
- Vacuum Assisted Birth: Birth by vacuum assist and exclusive breastfeeding at 3 months of age
- Gestational Diabetes: Birth afflicted by gestational diabetes and exclusive breastfeeding at 3 months of age
- Preeclampsia: Birth afflicted by preeclampsia and exclusive breastfeeding at 3 months of age

SUMMARY:
The goal of this observational study is to learn about the effects of birth practices such as cesarean section and vacuum assisted birth and diseases such as gestational diabetes and preeclampsia on exclusive breastfeeding. The main question it aims to answer is:

• Does cesarean section, vacuum assisted birth, gestational diabetes and preeclampsia affect exclusive breastfeeding three months after birth? Participants answer eight online survey questions. One survey is distributed before birth and the remaining seven surveys are distributed after birth at three, seven and four-teen days, as well as one, three, six and twelve months after birth.

ELIGIBILITY:
Inclusion Criteria: 18 years, intention to breastfeed, single gestation, reads and understands Danish -

Exclusion Criteria: Twin gestation, less than 18 years, no intention to breastfeed, does not read and understand Danish

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and women who have given birth > 18 years old
Sampling Method: Probability Sample
Enrollment: 1628 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Exclusive Breastfeeding | 3 months
  Infant receives mothers milk exclusively

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bergholt, Professor, PhD, MSc, Principal Investigator — Herlev & Gentofte Hospital
Locations (1):
- Herlev & Gentofte University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Not at this time.